CLINICAL TRIAL: NCT05507281
Title: Efficacy of Ultrasound-guided Erector Spinae Plane Block Versus Retrolaminar Block for Postoperative Analgesia in Patients Undergoing Thoracotomy
Brief Title: Ultrasound-guided Erector Spinae Plane Block Versus Retrolaminar Block for Postoperative Analgesia in Thoracotomy
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Tanta University (Other)
Responsible Party: Principal Investigator, Fatma Adel Momen Elshazly, Principal Investigator, Tanta University
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 34580/3/21
Record Dates: First submitted 2022-08-17; First posted 2022-08-18 (Actual); Last update posted 2022-08-29 (Actual); Status verified 2022-08

CONDITIONS: Postoperative Analgesia; Retrolaminar Block; Ultrasound-guided Erector Spinae Plane Block; Thoracotomy

STUDY DESIGN:
Intervention Model Description: Patients were randomly allocated into 3 equal groups (Control group, Ultrasound-guided Erector Spinae Plane Block group, Retrolaminar Block, 20 patients each) through sealed envelopes.
Who Masked: Participant, Outcomes Assessor
Masking Description: An anesthesiologist gave the block and outcomes were obtained by another one blinded to the study group. PHILIPS ultrasound machine and high frequency linear array probe with a frequency of 5-13 MHZ will be used.
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Control group (Sham Comparator): Patients received general anesthesia alone.
  Interventions: Procedure: Control
- Ultrasound-guided Erector Spinae Plane Block (Experimental): A 22-gauge needle is inserted at a puncture site lateral to the target spinous process using ultrasound imaging and advanced until contact is made with the transverse process. The local anesthetic agent will be injected between the transverse process and the erector spinae muscle using 20 ml (19ml bupivacaine 0.25% plus 1ml dexamethasone 4mg).
  Interventions: Procedure: Ultrasound-guided Erector Spinae Plane Block
- Retrolaminar Block (Experimental): A 22-gauge needle is inserted at a puncture site lateral to the target spinous process using ultrasound imaging and advanced caudally or cranially until it contacts the lamina. The local anesthetic agent will be injected on the lamina using 20 ml (19ml bupivacaine 0.25% plus 1ml dexamethasone 4mg).
  Interventions: Procedure: Retrolaminar Block

INTERVENTIONS:
Procedure: Ultrasound-guided Erector Spinae Plane Block — ultrasound-guided ipsilateral Erector Spinae Plane Block (20 ml (19ml bupivacaine 0.25% plus 1ml dexamethasone 4mg)).
  Arms: Ultrasound-guided Erector Spinae Plane Block
Procedure: Retrolaminar Block — ultrasound-guided ipsilateral Retrolaminar Block (20 ml (19ml bupivacaine 0.25% plus 1ml dexamethasone 4mg)).
  Arms: Retrolaminar Block
Procedure: Control — General anesthesia
  Arms: Control group

SUMMARY:
Comparing efficacy of Ultrasound-guided Erector Spinae Plane Block versus Retrolaminar Block for Postoperative Analgesia in Patients Undergoing Thoracotomy

DETAILED DESCRIPTION:
Thoracotomy is one of the most painful surgical procedures. The reported incidence of persistent pain after thoracic surgery (post thoracotomy pain syndrome) has been reported in 20%-70% of patients. Inadequately treated post thoracotomy pain can have several negative consequences. Therefore, pain relief is essential to facilitate coughing and deep breathing and to promote early mobilization.

Thoracic epidural analgesia and thoracic paravertebral block are strongly recommended techniques for managing post thoracotomy pain to reduce opioid use and the related adverse effects as hypoventilation, depression of cough reflex, nausea and vomiting. However, they can be technically challenging to perform and are associated with up to 15% failure rate in Thoracic epidural analgesia and potential risk of pneumothorax in thoracic paravertebral block.

Erector spinae plane block is a relatively novel ultrasound-guided regional technique. Its application in patients with chronic thoracic neuropathic pain and acute surgical pain has been described by Forero et al.

Retrolaminar block is an easy and safe analgesic technique. It has been reported to be satisfactory for post-operative analgesia after breast surgery.

To our knowledge there is no clinical studies, comparing the effectiveness of both blocks on postthoracotomy pain, has been reported.

ELIGIBILITY:
Inclusion Criteria:

* Adult patients aged 21-65 years old of both sexes.
* Patients were scheduled for elective thoracotomy.
* Their ASA physical status classification is II-III.

Exclusion Criteria:

* Patients' refusal.
* Local infection at the site of block.
* Coagulation abnormalities.
* Sever spinal deformity e.g. scoliosis.
* Known hypersensitivity to local anesthetics.
* Mental dysfunction and cognitive disorders.
* History of drug abuse and chronic analgesic use.

Ages: 21 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 60 (Actual)
Dates: Start 2021-08-01 (Actual); Primary Completion 2022-08-01 (Actual); Study Completion 2022-08-01 (Actual)

PRIMARY OUTCOMES:
Pain assessment | 24 hours postoperatively.
  The Numeric Pain Rating Scale is a valid and simple approach to pain assessment (0= no pain and 10= worst possible pain). Postoperative pain will be assessed at emergence and 2nd, 4th, 8th, 12th, 18th and 24th hour postoperatively.

SECONDARY OUTCOMES:
The time of first analgesic request | 24 hours postoperatively
  The time of first analgesic request. IV morphine sulphate 0.05 mg/kg will be administered as rescue analgesic if Numeric Pain Rating Scale is ≥ 4.
The total amount of morphine | 24 hours postoperatively
  The total amount of morphine consumption in the first 24 hours postoperatively.

CONTACTS AND LOCATIONS:
Locations (1):
- Tanta University, Tanta, Gharbia Governorate, Egypt